CLINICAL TRIAL: NCT00035568
Title: A Research Study to Assess the Mechanism By Which Glucovance, Metformin, and Glyburide Work To Control Glucose Levels In Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: CV138-062
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucovance; Metformin; Glyburide

INTERVENTIONS:
Drug: Glucovance (metformin HCl/glyburide)
Drug: or Metformin HCl alone
Drug: or Glyburide alone.

SUMMARY:
The purpose of this clinical research study is to support earlier observations that Glucovance controls glucose levels after a mean, and improves overall glucose control better than metformin or glyburide therapy alone in adults with type 2 diabetes.

ELIGIBILITY:
Adults 20-75 with a diagnosis of type 2 diabetes mellitus who are not adequately controlled with diet and exercise, and have an HbA1c greater than 6.7%

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-02; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Los Angeles, California
  - Local Institution, Chicago, Illinois
  - Local Institution, Indianapolis, Indiana
  - Local Institution, Brooklyn, New York
  - Local Institution, Rochester, New York
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Dallas, Texas
  - Local Institution, San Antonio, Texas

REFERENCES:
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595